CLINICAL TRIAL: NCT06554977
Title: Platelets to Albumin Ratio for Prediction of Acute Kidney Injury in Patients Admitted to the Intensive Care Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ola Mohammed Hussein Mohammed, Physician, Assiut University
Other Study IDs: Aki in icu patients
Record Dates: First submitted 2024-07-26; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Platelets/Albumin and Aki
MeSH Terms: interventions — Laboratories

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with Aki: acute kidney injury that will be divided into transient and persistent Aki according to follow up within 48hr and 72hr with kidney function (urea & creatine)
  Interventions: Other: Laboratory
- Non Aki patients
  Interventions: Other: Laboratory

INTERVENTIONS:
Other: Laboratory — CBC Kidney function (Urea, creatine) Platelets to albumin ratio Albumin /creatine ratio CRP Urine analysis Abdominal us Kidney function , CBC , Albumin will be done at the time of admission i

SUMMARY:
To evaluate the role of platelet to albumin ratio to detect Acute kidney injury in patients admitted to intensive care

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common clinical syndrome characterized by a sudden decline in or loss of kidney function. AKI is not only associated with substantial morbidity and mortality but also with increased risk of chronic kidney disease (CKD). AKI is classically defined and staged based on serum creatinine concentration and urine output rates. The etiology of AKI is conceptually classified into three general categories: prerenal, intrarenal, and postrenal Acute kidney injury (AKI) is a complex systemic syndrome associated with high morbidity and mortality. Among critically ill patients admitted to intensive care units (ICUs), the incidence of AKI is as high as 50% and is associated with dismal outcomes. Thus, the development and validation of clinical risk prediction tools that accurately identify patients at high risk for AKI in the ICU is of paramount importance Since the 2017 Acute Disease Quality Initiative (ADQI) workgroup proposed standard definitions of transient and persistent AKI (pAKI) based on the potential impact of AKI duration on outcomes numerous investigators explored the outcomes of different types of AKI. Previous evidence indicated that two-thirds of patients with AKI resolve their renal dysfunction rapidly and there still almost one-third of patients progress to pAKI. pAKI patients exhibited an increased risk of CKD, ESKD, prone to receive RRT, and reduced survival compared to those transient AKI patients Considering the important role of pAKI in the prognosis of critically ill patients, early and accurate risk assessment is of critical importance for clinical management in ICU patients to receive early interventions. Clinicians are seeking clinically meaningful predictors or biomarkers for pAKI in ICU patients. A recent study intended to assess novel candidate biomarkers to predict pAKI in critically ill patients and found that urinary C-C motif chemokine ligand 14 is a predictive biomarker for pAKI in critically ill patients Shen et al. reported that 24-h procalcitonin change is a good predictor of pAKI in critical patients However, these biomarkers are not easily obtained upon admission to clinical. A simple and easily accessible prognostic biomarker for early risk stratification of pAKI in patients admitted to ICU is needed. Platelet to albumin ratio (PAR) is a widely used biomarker clinically based on routine laboratory tests which reflect the systemic inflammatory state and nutrition status, has been reported to predict several disease settings

ELIGIBILITY:
Inclusion Criteria:

* (1) Patient admitted to ICU whatever the cause ( 2) KDIGO-AKI criteria based on serum creatinine in the first 48 h of their ICU. admission

Exclusion Criteria:

* less than 18-year-old at first admission to ICU; (3) more than 10% of personal data was missing; (4) patients with repeated ICU admissions; (5) patients without serum creatinine measures between 48 and 72 h after the diagnosis of AKI (6) pregnant women . (7) patient known chronic kidney disease. (8) Patient with End stage renal disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to icu number of patients 140
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Detect relation between platelets to albumin ratio for prediction of transient or persistent AKI in ICU patients | 2years
  T he included patients will be divided into two groups according to the optimal cut-off value of
  PAR: high-PAR group (≥ 7.2), low-PAR group (< 7.2). Number of patients is 140

SECONDARY OUTCOMES:
Effect of the cause of ICU admission on platelets to albumin ratio and persistent AKI | 2years
  - Relation between platelets to albumin ratio to hospital stay 2- Relation of platelets to albumin ratio to the need for ranel replacement therapy